CLINICAL TRIAL: NCT00179582
Title: A Randomized, Multi-center, Double-blind, Placebo Controlled, Dose Ranging Study With VSL#3 in Diarrhea Predominant IBS Patients
Brief Title: Dose Ranging Study With the Probiotic Combination (VSL#3) in Diarrhea IBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Lembo, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004P000001; VSL1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: IBS
Keywords: IBS; Functional bowel disorder; Diarrhea; probiotic
MeSH Terms: conditions — Diarrhea

INTERVENTIONS:
Drug: VSL#3

SUMMARY:
To evaluate the effects of VSL#3 on symptoms associated with diarrhea predominant IBS

DETAILED DESCRIPTION:
The study will evaluate 2 doses of VSL#3 and placebo over a 4 week period in patients presenting with diarrhea predominant IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* IBS diarrhea

Exclusion Criteria:

* < 18 years of age
* Pregnancy/breast feeding
* concomitant medications to reduce bowel function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Global improvement in IBS symptoms

SECONDARY OUTCOMES:
Frequency of bowel movements
Changes in abdominal pain
Changes in bloating

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lembo, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- BIDMC, Boston, Massachusetts, United States

REFERENCES:
- [Result] Niv E, Naftali T, Hallak R, Vaisman N. The efficacy of Lactobacillus reuteri ATCC 55730 in the treatment of patients with irritable bowel syndrome--a double blind, placebo-controlled, randomized study. Clin Nutr. 2005 Dec;24(6):925-31. doi: 10.1016/j.clnu.2005.06.001. Epub 2005 Jul 27. PMID 16051399